CLINICAL TRIAL: NCT04998149
Title: The Effect of the Use of a Peanut Ball on Labor Time and "Pushing" After Epidural Anesthesia in Nulliparous Women.
Brief Title: The Effect of the Use of Peanut Ball on Labor Time in Nulliparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Ani Jacob, Nurse Scientist, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-0330
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Laboring Women

STUDY DESIGN:
Intervention Model Description: There will be a standard group and an intervention group selected by BRMS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- standard care (No Intervention): The control group subjects will receive standard of care during labor using pillows and wedges as positional devices.
- Peanut ball intervention (Experimental): The experimental group will receive peanut ball as positioning device during labor
  Interventions: Device: Peanut Ball positioning device

INTERVENTIONS:
Device: Peanut Ball positioning device — Peanut Ball manufactured by Clinton industries at graylinemedical.com https://www.graylinemedical.com/products/clinton-industries-peanut-ball-peanut-ball-40-cm-yellow-8540?_pos=3&_sid=d6e52e63c&_ss=r
  Arms: Peanut ball intervention

SUMMARY:
Peanut ball use has become popular with midwives and nurses because it is an inexpensive, nonpharmacological intervention that can help with positioning the patient to decrease labor time. The peanut ball allows the patient to reposition her legs in a way that mimics squatting and changes the diameter of the pelvis. This can aid in cervical dilatation and the descent of the fetus. In turn, laboring down can decrease the time spent pushing and prevent maternal exhaustion.

This study aims to test the following hypotheses:

The use of the peanut ball compared to standard of care will:

1. Reduce the time (in minutes) between administration of epidural and complete cervical dilation
2. Reduce pushing time as measured by duration of time pushing to the delivery of the baby
3. Decrease the rate of cesarean sections in nulliparous women

DETAILED DESCRIPTION:
This is a randomized control study. Each patient who meets the inclusion criteria will be informed about the study within 12 hours of admission to the unit. When the participant is alert and prior to administration of medicinal pain relief measures, the patient will be asked to consent to be a participant. Basic admission demographic information will be collected from the electronic medical record (EMR) and will be used to identify potential subjects (inclusion/exclusion criteria). Recruitment will include a scripted informative conversation with the potential subject along with an informed consent to further determine eligibility and willingness to participate in the study.

The peanut ball size will be determined by the patient weight indicated on the peanut ball itself and compared with the patient's documented weight in the EMR. The ball will be inflated prior to use and a pictorial introduction of how to use the peanut ball will be shown to the study subject.

The peanut ball use will be discontinued immediately prior to the delivery of the baby. The study time will be documented and calculated for all subjects (treatment and control) from the time of introduction of epidural analgesia to the delivery of the baby.

The proposed Peanut Ball manufactured by Clinton industries at graylinemedical.com is made from durable, ribbed, heavy-walled, polyvinyl chloride (PVC) material, burst resistant, deflate slowly if punctured, and latex free with non-slip grip ridges. It is available in variable sizes ranging from 40 cm-70 cm in length. It is re-usable, after cleaning with hospital grade wipes. It is recommended that the peanut balls should be protected from sunlight and sharp objects.

ELIGIBILITY:
Inclusion Criteria:

Women between 18 -50 years of age presenting in labor or for induction of labor

* Nulliparous (first delivery)
* 37 0/7- 41 6/7 weeks of gestation
* Singleton, Vertex presentation
* Plan to deliver with epidural anesthesia
* Has had at least one vaginal exam to determine the cervical dilatation prior to the proposed intervention
* Prescribed Oxytocin (Pitocin)

Exclusion Criteria:

* Multi gravida women
* Admitted in second stage of labor
* Multiple gestations
* Non-vertex presentations
* Women receiving magnesium sulfate
* Preterm or post term labor (<37 weeks or >42 weeks)
* Women with hypertensive disorders of pregnancy
* Diabetes including gestational diabetes
* Muscular or skeletal limitations that does not allow for positioning
* Un-medicated labors ( delivery without epidural, about 5-20% )
* Category III fetal heart rate tracings
* Suspected infections (e.g. STDs, viral/bacterial infections)
* Planned cesarean delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Decrease labor time | From epidural analgesia to delivery of the baby
  The primary outcome goal is to decrease the length of first and second stage of labor in nulliparous women after receiving epidural analgesia, measured in minutes

SECONDARY OUTCOMES:
Decrease cesarean section deliveries | From epidural analgesia to delivery of the baby
  to decrease the rate of cesarean births among nulliparous women and to decrease the rate of operative vaginal deliveries (forceps/vacuum) by 10%.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Huntington Hospital, Huntington, New York
  - North Shore University Hospital, Manhasset, New York
  - Northwell health, Northern Westchester Hospital, Mount Kisco, New York
  - Northwell Health, Peconic Bay Medical Center, Riverhead, New York

IPD SHARING:
Plan to Share IPD: No
Only aggregated study results/data will be shared with other researchers. Individual participant data will not be shared.

REFERENCES:
- [Background] Delgado A, Maia T, Melo RS, Lemos A. Birth ball use for women in labor: A systematic review and meta-analysis. Complement Ther Clin Pract. 2019 May;35:92-101. doi: 10.1016/j.ctcp.2019.01.015. Epub 2019 Feb 2. PMID 31003693
- [Background] Tussey CM, Botsios E, Gerkin RD, Kelly LA, Gamez J, Mensik J. Reducing Length of Labor and Cesarean Surgery Rate Using a Peanut Ball for Women Laboring With an Epidural. J Perinat Educ. 2015;24(1):16-24. doi: 10.1891/1058-1243.24.1.16. PMID 26937158
- [Background] Randomized Controlled Trial of Use of the Peanut Ball During Labor. MCN Am J Matern Child Nurs. 2016 May-Jun;41(3):E9-E10. doi: 10.1097/NMC.0000000000000240. No abstract available. PMID 27128653